CLINICAL TRIAL: NCT00261404
Title: A Phase II, Open Label, Single Arm, "Proof of Concept" Study of TNFerade™ Plus Radiation in Patients With Metastatic Melanoma
Brief Title: TNFerade™ Biologic Plus Radiation for Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Other Study IDs: GV-001.008
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Drug: TNFerade™

SUMMARY:
Phase II, open label study in which patients with metastatic melanoma (stage III or IV) who have cancer which is not considered curable by surgery will receive intratumoral injections of TNFerade™ plus radiation as a 4-week treatment, followed by a 3 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years old or older, and able to give informed consent.
* Patients with metastatic melanoma (AJCC stage III or IV) who are not eligible for curative surgery and who are candidates for experimental therapy. Eligible patients will include those with melanoma involving the regional lymph nodes and surrounding tissues as well as those with unresectable cutaneous, subcutaneous, nodal or soft tissue metastases.
* Patients must have one or more tumor nodules accessible for direct injection.
* Patients with metastases outside the treatment field may be enrolled if the sites of metastases do not limit survival expectancy to less than 3 months.
* Patients must be unlikely to derive significant potential benefit from other treatment options and no other treatments should be anticipated during the study treatment period or a period of two months thereafter.
* Patient's Karnofsky performance status must be greater than or equal to 70%.

Exclusion Criteria:

* Chemotherapy or experimental medications within the last four weeks prior to Day 1.
* Active disease of the central nervous system.
* Baseline liver enzymes (AST, ALT, bilirubin, alkaline phosphatase) greater than 3 times the upper limit normal.
* Renal insufficiency (Serum creatinine greater than 2.0 mg/dL).
* Coagulopathy (PT INR >1.5 or PTT ratio >1.5 in patients not receiving anticoagulants).
* Significant anemia (e.g. hematocrit <28% or hemoglobin <9 g/dL). May have RBC transfusion, or thrombocytopenia (platelet count less than 100,000/μl); or leukopenia (WBC <3000/μl; ANC <1500/μl).
* Patients with documented history of deep venous thrombosis, pulmonary embolus, cerebrovascular disease, stroke, or TIA.
* Patients with history of coagulopathy or known thrombophillic disorders.
* Clinical evidence of active infection of any type, including hepatitis B or C virus.
* Pregnant or lactating women. It is recommended that both men and women use condoms or another barrier method of birth control for at least 2 months following the last administration of TNFerade™ biologic and some form of birth control for at least 1 year.
* Significant concurrent medical or psychiatric illness which, in the opinion of the investigator, would interfere with the patient's ability to participate in the trial
* Chronic systemic corticosteroid use, orally or parenterally administered.
* Known sensitivity to lidocaine, procaine or amide local anesthetics (used for topical anesthesia).
* Surgery within the last 4 weeks prior to day 1 (if patient was ambulatory within 48 hours of surgery, patient may be considered eligible)
* Attempted resection of the tumor to be treated, or surgery on the area to be treated, with incomplete healing of surgical wound. (If the surgical wounds are completely healed and lesion continues to progress, patient may be enrolled.)
* Patients with a history of clinical lymphedema in the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Crowley Medical Research Center, Dallas, Texas, United States